CLINICAL TRIAL: NCT02175030
Title: RAPID EC - Randomized Controlled Trial Assessing Pregnancy With Intrauterine Devices for Emergency Contraception
Brief Title: RAPID EC - Rct Assessing Pregnancy With Intrauterine Devices for EC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, David Turok, M.D., University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 73554
Record Dates: First submitted 2014-06-23; First posted 2014-06-26 (Estimated); Results first posted 2022-06-29 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Contraception
Keywords: Emergency contraception; Levonorgestrel IUD; Copper IUD
MeSH Terms: interventions — Intrauterine Devices, Copper

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Copper T380 IUD (Active Comparator): Randomized to copper T380 IUD for EC (emergency contraception)
  Interventions: Drug: Copper IUD
- LNG20 IUD (Active Comparator): Randomized to LNG20 IUD for EC (emergency contraception)
  Interventions: Drug: Levonorgestrel IUD

INTERVENTIONS:
Drug: Copper IUD — Randomization to copper/Paragard IUD for emergency contraception
  Other Names: Paragard IUD
  Arms: Copper T380 IUD
Drug: Levonorgestrel IUD — Randomization to Levonorgestrel/Mirena IUD for emergency contraception
  Other Names: Mirena IUD, LNG20 IUD, Levonorgestrel IUD, Liletta IUD
  Arms: LNG20 IUD

SUMMARY:
This study is a randomized trial of two IUDs for emergency contraception: the copper IUD, the most effective method of emergency contraception vs. the levonorgestrel IUD, the most preferred IUD which has never been tested as an emergency contraceptive. This research has the potential to increase use of highly effective contraception in a high-risk population and lower the persistently elevated rate of U.S. unintended pregnancy.

DETAILED DESCRIPTION:
Unintended pregnancy has multiple adverse effects on both maternal and child health. The United States continues to have one of the highest rates of unintended pregnancy among developed countries. To combat this problem, we are studying initiation of the highly effective intrauterine device (IUD) for women presenting for emergency contraception (EC). This is an ideal population to initiate highly effective reversible contraception (HERC) as they are at high risk of unintended pregnancy and are acting to reduce that risk. We have recently demonstrated significantly lower pregnancy rates 12 months after presenting for EC among women who selected the copper IUD versus those who selected oral Levonorgestrel (LNG).

Not only is the copper IUD the most effective method of EC, it is considered a top tier anticipatory contraception method and its ability to prevent pregnancy is on par with tubal sterilization (less than 1% in the first year with lower failure rates in subsequent years). However, women selecting intrauterine contraception have shown a strong preference for the LNG IUD. The LNG IUD, is as effective at preventing pregnancy as the Copper IUD, and has some non-contraceptive effects that many women see as benefits such as the reduction or elimination of menstrual bleeding and menstrual related discomfort. Of currently available reversible contraceptives, the LNG IUD has the highest levels of user satisfaction and continuation. However, its effectiveness as an emergency contraceptive remains unknown. A randomized control trial is necessary to assess the safety and efficacy of the LNG IUD as EC. Demonstrating the efficacy, safety, and acceptability of the LNG IUD for EC will improve options for women seeking EC and who desire a highly effective method of contraception.

ELIGIBILITY:
Inclusion Criteria:

* Females between 18-35 years old
* In need of EC (had unprotected intercourse within 120 hours - 5 days)
* Desire to prevent pregnancy for 1 year
* Fluent in English and/or Spanish
* Have a regular menstrual cycle (21-35 days)
* Know their last menstrual period (+/-3 days)
* Be willing to comply with the study requirements
* Desire to initiate an IUD
* Negative urine pregnancy test

Exclusion Criteria:

* Current pregnancy
* Breastfeeding
* Intrauterine infection within the past three months
* Sterilization
* Already have an IUD or contraception implant (Nexplanon) in place
* Vaginal bleeding of unknown etiology
* Known Gonorrhea or Chlamydia infection in the last 30 days (unless successfully treated at least 7 days prior to study entry)
* Known abnormalities of the uterus that distort the uterine cavity
* Allergy to copper
* Use of oral Emergency Contraception in the preceeding 5 days

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 711 (Actual)
Dates: Start 2016-08; Primary Completion 2020-02 (Actual); Study Completion 2020-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Turok, MD, Principal Investigator — University of Utah
Locations (6):
- United States (6):
  - Planned Parenthood Association of Utah, Logan, Utah
  - Planned Parenthood Association of Utah, Ogden, Utah
  - Planned Parenthood Association of Utah, Orem, Utah
  - Planned Parenthood Association of Utah, Salt Lake City, Utah
  - Planned Parenthood Association of Utah, South Jordan, Utah
  - Planned Parenthood Association of Utah, West Valley City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kaiser JE, Turok DK, Gero A, Gawron LM, Simmons RG, Sanders JN. One-year pregnancy and continuation rates after placement of levonorgestrel or copper intrauterine devices for emergency contraception: a randomized controlled trial. Am J Obstet Gynecol. 2023 Apr;228(4):438.e1-438.e10. doi: 10.1016/j.ajog.2022.11.1296. Epub 2022 Nov 23. PMID 36427600
- [Derived] BakenRa A, Gero A, Sanders J, Simmons R, Fay K, Turok DK. Pregnancy Risk by Frequency and Timing of Unprotected Intercourse Before Intrauterine Device Placement for Emergency Contraception. Obstet Gynecol. 2021 Jul 1;138(1):79-84. doi: 10.1097/AOG.0000000000004433. PMID 34259467
- [Derived] Boraas CM, Sanders JN, Schwarz EB, Thompson I, Turok DK. Risk of Pregnancy With Levonorgestrel-Releasing Intrauterine System Placement 6-14 Days After Unprotected Sexual Intercourse. Obstet Gynecol. 2021 Apr 1;137(4):623-625. doi: 10.1097/AOG.0000000000004118. PMID 33706343
- [Derived] Turok DK, Gero A, Simmons RG, Kaiser JE, Stoddard GJ, Sexsmith CD, Gawron LM, Sanders JN. Levonorgestrel vs. Copper Intrauterine Devices for Emergency Contraception. N Engl J Med. 2021 Jan 28;384(4):335-344. doi: 10.1056/NEJMoa2022141. PMID 33503342

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Copper T380 IUD | LNG20 IUD
Started | 356 | 355
Completed | 321 | 317
Not Completed | 35 | 38
Not completed — Failed screen after consent | 7 | 6
Not completed — Failed IUD Insertion | 20 | 21
Not completed — Physician Decision | 1 | 1
Not completed — Lost to Follow-up | 6 | 6
Not completed — Withdrawal by Subject | 1 | 4

BASELINE CHARACTERISTICS:
Population: Participants randomized to receive either the Copper T380 IUD or LNG20 IUD as emergency contraception
Groups:
- Total: Total of all reporting groups
Arm/Group | Copper T380 IUD | LNG20 IUD | Total
Number analyzed (Participants) | 328 | 327 | 655
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 328 | 327 | 655
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.9 (4.6) | 24.0 (4.9) | 24.0 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 328 | 327 | 655
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 182 | 171 | 353
  Hispanic / Latina | 101 | 111 | 212
  Asian | 11 | 11 | 22
  Native Hawaiian / Pacific Islander | 8 | 5 | 13
  American Indian / Alaska Native | 10 | 10 | 20
  Black / African American | 12 | 12 | 24
  More than one race | 4 | 7 | 11
Region of Enrollment [Number; unit: participants]
  United States | 328 | 327 | 655

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Reporting a Pregnancy
Description: Urine pregnancy tests within 30 days after IUD insertion will be performed either at home or in clinic. We will use the total number of pregnancies per ARM and the overall number of participants analyzed per ARM to calculate, for each ARM, the percentage of participants reporting a pregnancy in the first month of use of the IUD.
Time Frame: 1 month after enrollment
Population: Urine pregnancy tests within 30 days after IUD insertion will be performed either at home or in clinic.
Measure: Number (95% Confidence Interval); unit: % of participants reporting pregnancy
Arm/Group | Copper T380 IUD | LNG20 IUD
Number analyzed (Participants) | 321 | 317
% of participants reporting pregnancy | 0 [0 to 1.1] | 0.3 [0.01 to 1.7]

2. Secondary Outcome: Number of Participants With Unintended Pregnancy After Initiating the Levonorgestrel IUD Versus the Copper T380 IUD for EC at One Year.
Description: Participants will be followed for pregnancies at regular intervals throughout the year and pregnancies will be recorded.
Time Frame: 1 year after enrollment
Population: This denominator excludes participants lost to follow-up and participants who cited a desire for pregnancy as their reason for removing their IUD, but includes all other participants who removed their IUD throughout the 12 months follow-up and all participants with an expelled IUD.
Measure: Count of Participants; unit: Participants
Arm/Group | Copper T380 IUD | LNG20 IUD
Number analyzed (Participants) | 313 | 315
Participants | 7 | 7

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during the year of follow-up collectively and defined as all events requiring additional medical care in the first month of use of IUD.
Description: Definition of adverse events does not differ from definition used by clinical trials.gov.
  Adverse events were collected as part of routine follow-up surveys completed by participants and reviewed by PI for determination of Serious Adverse Event collectively and reported collectively as all events requiring additional medical care in the first month of use after IUD insertion.
Arm/Group | Copper T380 IUD | LNG20 IUD
All-Cause Mortality (participants affected / at risk) | 0/328 | 0/327
Serious Adverse Events (participants affected / at risk) | 0/328 | 0/327
Other Adverse Events (participants affected / at risk) | 16/328 | 17/327
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Copper T380 IUD (N=328) | LNG20 IUD (N=327)
Adverse events experienced related to IUD at 1-Month (Reproductive system and breast disorders) | 16 (16) | 17 (17)

LIMITATIONS AND CAVEATS:
This was a randomized trial. Implications for clinical care may vary when people choose their treatment options.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-10): https://cdn.clinicaltrials.gov/large-docs/30/NCT02175030/Prot_SAP_000.pdf
  • Informed Consent Form (2019-11-26): https://cdn.clinicaltrials.gov/large-docs/30/NCT02175030/ICF_001.pdf